CLINICAL TRIAL: NCT01252992
Title: Paradoxical Reactions During Anti-mycobacterial Treatment of Extrapulmonary Tuberculosis in Non Immuno-compromized Patients : Clinical, Radiological et Immunological
Brief Title: Paradoxical Reactions in Non Immuno-compromized Patients With Extrapulmonary Tuberculosis
Acronym: PARATB
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P081253; 2010-A00375-34 (Other: ID-RCB)
Record Dates: First submitted 2010-11-27; First posted 2010-12-03 (Estimated); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Extrapulmonary Tuberculosis
Keywords: Extrapulmonary; Tuberculosis; Paradoxical reaction; Risk factors; Incidence; CT scan; Natural history; Immune system phenomena; Immune markers; Gene Expression Profiling
MeSH Terms: conditions — Tuberculosis, Extrapulmonary; Tuberculosis | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (immunologic test), DNA, RNA, Biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1:paradoxical reaction negative (RP-): control group with tuberculosis but without paradoxical reaction
  Interventions: Genetic: Genetic analysis; Radiation: Body scan (CERVICO THORACO ABDOMINAL) + Cranian IRM; Other: Immunologic analysis
- 1:paradoxical reaction negative (RP+): group with tuberculosis and paradoxical reaction
  Interventions: Genetic: Genetic analysis; Radiation: Body scan (CERVICO THORACO ABDOMINAL) + Cranian IRM; Other: Immunologic analysis; Other: QuantiferonTB Gold test

INTERVENTIONS:
Genetic: Genetic analysis — 1. identification of candidates genes by a differential analysis of the whole transcriptome of the peripheral leucocytes of 20 PR+ patients and 20 RP- controls, at D0, D15, M2,;
  2. Genetic association analysis: comparison of allelic distributions of SNPs (diallelic markers) within the candidate genes, between PR+ and PR- patients, in the whole cohort.
  One supplementary ACD tube of 5 ml à D0, D15, M2, PR+, for RNA extraction.
Radiation: Body scan (CERVICO THORACO ABDOMINAL) + Cranian IRM — at day 0, Month 2, paradoxical reaction, end of treatment, read by an independent radiologist
Other: Immunologic analysis — For patients included until 20 PR+ : blood puncture of 4 ACD tubes of 10 ml, 1 EDTA tube of 7,5 ml et 1 heparinate lithium tube of 7,5ml at D0, D15, M2, and M6 and at the time of an potential RP+
Other: QuantiferonTB Gold test — at M0, M2, M6 and in case of PR+.
  Groups: 1:paradoxical reaction negative (RP+)

SUMMARY:
Tuberculous paradoxical reactions (PR) are immune reactions occurring during the course of antituberculous treatment and leading to a worsening of tuberculous symptoms after an initial improvement. This phenomenon has very extensively studied in HIV infected patients where it corresponds to the so called IRIS (immune reconstitution syndrome). However, it laso occurs in non immuno-compromized patients, especially those with extra-pulmonary localization of tuberculosis. The aim of the study is to look for risk factors of paradoxical reaction in non immuno-compromized patients with extra-pulmonary tuberculosis. The investigators will consider clinical, radiological and biological variables, including specific immune and genetic markers. Our secondary goals are to estimate the incidence of PR, describe their natural history; characterize the type of immune response they correspond to, and look for better diagnostic tools.The immunological characterization and the finding of predictive factors of PR, especially the genetic ones will allow a better understanding of biological mechanisms that lead to their occurrence during extra-pulmonary tuberculosis treatment. The establishment of predictive criteria could permit a better surveillance of at risk patients for a rapid treatment, or even a prevention of PR. The establishment of new diagnostic criteria at the time of PR could avoid numerous invasive diagnostic procedures, surgery and/or useless prolongation of antibiotic treatment.

DETAILED DESCRIPTION:
Primary objective :

Search for predictive factors of tuberculous paradoxical reaction (PR), with assessment of clinical, radiological and biological factors.

Secondary objectives :

* Descriptive study of PR : incidence, clinical and radiological presentation, clinical course ; characterization of mycobacteria strains- Search for genetic predictive factors of PR
* Characterization of the specific immune antigene response during PR et analysis of different cell subsets implicated in peripheral blood and locally- Characterization of the anti-bacterial immune response before and after antituberculous treatment
* Preliminary search for new diagnosis criteria including clinical, biological (immune and genetic) and radiological factors.Methodology : Multicentric cohort study for a total of 5 years (4 years of enrolment and one year of follow-up, with biological collection for scientific purpose

Inclusion Status of patients (determined by a validation comity at M6)

* PR+ : PR with clinical symptoms
* rPR : pure radiological PR
* PR- : absence of RP after 6 months of treatment Development of the study

Primary outcome :

- Association between PR+ occurrence and clinical, biological and radiological factors harvested at the diagnosis of tuberculosis..

Secondary outcomes :

* Association between PR+ and rPR
* occurrence and the above quoted factors.- Descriptive study : clinical, biological, and radiological presentation of PR+ and rPR, characterization of isolated BK strains in PR+ patients
* Immunological study in 20 PR+ patients and 20 RP- : 20 patients per group will allow a 80% power to detect, by means of bilateral Mann-Whitney test with alpha=5%, any difference in the count of specific cells corresponding to at least one standard deviation of the primary immunological outcome
* controls: variation between tuberculosis diagnostic and either PR time or M2 (in absence of PR), of the specific cells, macrophages, dendritic cells, gamma-delta lymphocytes, NK et CD4 cells counts
* Preliminary search for diagnostic criteria that can be used at the time of PR occurrence: variation between D0 and the PR of clinical, biological, radiological immunological et genomic of PR+ patients.
* Evolution specific and non specific immune response of mycobacterial antigen at tuberculosis diagnosis during tuberculosis treatment and after. Sample size calculation
* prognostic study : Patients will be recruited and followed until the achievement of a 20 PR+ sample. The investigators will have to analyze 200 patients.

ELIGIBILITY:
Inclusion Criteria:

* Extrapulmonary tuberculosis, with associated pulmonary localization or not
* Treatment started less than 5 days ago
* Negative HIV serology
* Social insurance
* Age >= 18- Foreseeable follow-up of at last one year
* Signed Free Inform Consent

Exclusion Criteria:

* HIV infection
* immuno-suppressive treatment (including corticosteroids > 10 mg /d prednisone equivalent, however patients with corticotherapy could be included during the phase 2 of the study)
* central neurological system tuberculosis and tuberculous pericarditis - pure pulmonary tuberculosis
* multiresistant tuberculosis
* pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Extra-pulmonary tuberculosis
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2011-03-14 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
Risk factors of paradoxical reaction | at 6 months
  Risk factors of paradoxical reaction : clinical, radiological immune and genetic factors

SECONDARY OUTCOMES:
Incidence and natural history of paradoxical reactions | during the first 6 months
Immune description of paradoxical reactions | during the first 6 months
Preliminary study of Diagnosis factors of paradoxical reaction | during the first 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne BOURGARIT, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Georges Pompidou Hospital, Paris, France